CLINICAL TRIAL: NCT01091857
Title: Mediators and Moderators of Exercise Behavior Change
Acronym: COSTRIDE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Other
Other Study IDs: 0604.12; 1R01CA109858-01 (NIH)
Record Dates: First submitted 2010-03-22; First posted 2010-03-24 (Estimated); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Validate STRIDE Exercise Intervention in Sedentary Individuals; Increase Positive Attitudes, Perceived Normative Support, Self-efficacy, and Intentions; Increase Self-reported Physical Activity
Keywords: Exercise; Transdisciplinary; Physiology; Mood; Motivation
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise intervention (STRIDE) (Experimental)
  Interventions: Behavioral: STRIDE
- Health and Wellness Control (Active Comparator)
  Interventions: Behavioral: STRIDE

INTERVENTIONS:
Behavioral: STRIDE

SUMMARY:
Rates of cancer and cardiovascular disease have shown very little improvement over the past two decades, and the incidence of Type II diabetes mellitus is increasing at an alarming rate. Recent reports estimate that approximately 30% of total cancer deaths are related to poor exercise and nutrition, and other reports have suggested that, when taking into consideration both cardiovascular disease and cancer, inactivity contributes to as many as 250,000 premature deaths per year (Booth et al., 2002). Despite the benefit of regular physical activity in the prevention of cancer and other debilitating illnesses, 75% of the U.S. population do not get the recommended amount of physical activity as defined by 30 minutes of moderate intensity physical activity 5 or more days per week (CDC, 2001), and 40% of the population is completely sedentary (USDHHS, 19960. The objective of the proposed research is to understand the mediators and moderators of a well-tested individually tailored, print-based intervention to increase exercise behavior among sedentary adults. Using a randomized, controlled intervention ton trial, the proposed study will address three primary and one secondary hypotheses: 1) A previously tested and validated exercise promotion intervention (c.f., Marcus et al., 1998) is successful at helping sedentary individuals initiate and maintain a moderate intensity physical activity regimen, as compared to a health and wellness control intervention, 2) Increases in positive attitudes, perceived normative support, self-efficacy, and intentions to exercise will mediate the effectiveness of the intervention, 3) That increased positive mood, and better temperature, stress, and lactate regulation immediately after exercise challenge (assessed in the laboratory) will moderate the effectiveness of the intervention, and 4) Secondarily, we will test whether gender, race/ethnicity, and two recently suggested genetic factors (BDNF and OPRM1) moderate the effectiveness of the intervention. The rigorous assessment of how and for whom an exercise promotion intervention is effective will provide information for future development of intervention strategies and content, as well as allow the targeting of exercise content to individuals for whom it is most likely to be effective.

ELIGIBILITY:
Inclusion Criteria:

* All participants were required to exercise less than 90 minutes per week on average, have a body mass index (BMI) between 18 and 37.5, be physically capable of engaging in moderate-intensity physical activity, have a regular menstrual cycle (if female), be willing to be randomly chosen for one of the two interventions, and give informed consent.

Exclusion Criteria:

* Individuals were excluded if they smoked cigarettes, were on a restricted diet, taking psychotropic medications, receiving treatment for any psychiatric disorder, diabetic, had a history of cardiovascular or respiratory disease, had the flu or illness in the previous month, or were pregnant (if female).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 238 (Actual)
Dates: Start 2004-09; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Self-reported physical activity | 3,6,9,and 12 months post baseline
  After being randomly assigned to the exercise or health-and-wellness conditions, participants were followed up every three months for one year at which times they reported their current physical activity.

CONTACTS AND LOCATIONS:
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States

REFERENCES:
- [Derived] Bryan AD, Magnan RE, Hooper AE, Ciccolo JT, Marcus B, Hutchison KE. Colorado stride (COSTRIDE): testing genetic and physiological moderators of response to an intervention to increase physical activity. Int J Behav Nutr Phys Act. 2013 Dec 21;10:139. doi: 10.1186/1479-5868-10-139. PMID 24359456
- [Derived] Magnan RE, Kwan BM, Bryan AD. Effects of current physical activity on affective response to exercise: physical and social-cognitive mechanisms. Psychol Health. 2013;28(4):418-33. doi: 10.1080/08870446.2012.733704. Epub 2012 Oct 23. PMID 23088712
- [Derived] Magnan RE, Kwan BM, Ciccolo JT, Gurney B, Mermier CM, Bryan AD. Aerobic capacity testing with inactive individuals: the role of subjective experience. J Phys Act Health. 2013 Feb;10(2):271-9. doi: 10.1123/jpah.10.2.271. Epub 2012 Feb 29. PMID 22398432